CLINICAL TRIAL: NCT00537810
Title: Treatment of Binge Eating in Obese Patients in Primary Care
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Carlos Grilo, Professor of Psychiatry, Yale University
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0501027352; R01DK073542-01A1 (NIH)
Record Dates: First submitted 2007-09-27; First posted 2007-10-01 (Estimated); Results first posted 2014-12-12 (Estimated); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Obesity; Binge Eating
Keywords: Obesity; Binge eating; Sibutramine; Self-help; Primary care
MeSH Terms: conditions — Obesity; Bulimia | interventions — sibutramine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Sibutramine (Experimental): Sibutramine 15 mg daily
  Interventions: Drug: Sibutramine
- Placebo (Placebo Comparator): Placebo Daily
  Interventions: Drug: Placebo
- Placebo/CBTsh (Experimental): Placebo and Self-help CBT Placebo daily, Cognitive behavioral self-help manual for binge eating
  Interventions: Behavioral: Self-help CBT + Sibutramine
- Sibutramine/CBTsh (Experimental): Sibutramine and Self-help CBT 15 mg daily Cognitive behavioral treatment manual for binge eating
  Interventions: Behavioral: Self-help CBT + Placebo

INTERVENTIONS:
Drug: Sibutramine — 15 mg daily
  Other Names: Meridia
  Arms: Sibutramine
Drug: Placebo — Daily
  Arms: Placebo
Behavioral: Self-help CBT + Sibutramine — Cognitive behavioral treatment manual for binge eating Sibutramine 15 mg daily
  Arms: Placebo/CBTsh
Behavioral: Self-help CBT + Placebo — Cognitive behavioral treatment manual for binge eating Placebo daily
  Arms: Sibutramine/CBTsh

SUMMARY:
This study will test the effectiveness of two empirically-supported but distinct treatments for recurrent binge eating in obese patients: 1) Cognitive Behavior Therapy, using a pure self-help approach and 2) sibutramine, an anti-obesity medication also found to have efficacy for binge eating. Self-help Cognitive Behavior Therapy and sibutramine will be administered alone and in combination in a primary care setting.

ELIGIBILITY:
Inclusion Criteria:

* Obese (BMI >= 30)

Exclusion Criteria:

* Medication regimen that represents medical contraindication to sibutramine
* Serious unstable or uncontrolled medical conditions that represent contraindication to sibutramine
* Pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 104 (Actual)
Dates: Start 2007-09; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos M. Grilo, PhD, Principal Investigator — Yale University
Locations (3):
- United States (3):
  - Yale Internal Medicine Associates (YIMA), New Haven, Connecticut
  - Yale-New Haven Hospital (YNHH) Primary Care Center (PCC), New Haven, Connecticut
  - Yale Psychiatric Research at Congress Place, New Haven, Connecticut

REFERENCES:
- [Result] Grilo CM, Masheb RM, White MA, Gueorguieva R, Barnes RD, Walsh BT, McKenzie KC, Genao I, Garcia R. Treatment of binge eating disorder in racially and ethnically diverse obese patients in primary care: randomized placebo-controlled clinical trial of self-help and medication. Behav Res Ther. 2014 Jul;58:1-9. doi: 10.1016/j.brat.2014.04.002. Epub 2014 May 2. PMID 24857821
- [Derived] Correction to Grilo et al. (2015). J Consult Clin Psychol. 2015 Aug;83(4):747. doi: 10.1037/ccp0000043. PMID 26214545
- [Derived] Grilo CM, White MA, Masheb RM, Gueorguieva R. Predicting meaningful outcomes to medication and self-help treatments for binge-eating disorder in primary care: The significance of early rapid response. J Consult Clin Psychol. 2015 Apr;83(2):387-94. doi: 10.1037/a0038635. Epub 2015 Jan 26. PMID 25622201

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sibutramine | Placebo | Placebo/CBTsh | Sibutramine/CBTsh
Started | 26 | 27 | 25 | 26
Completed | 20 | 14 | 21 | 22
Not Completed | 6 | 13 | 4 | 4
Not completed — Withdrawal by Subject | 4 | 11 | 4 | 3
Not completed — Medically withdrawn | 2 | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sibutramine | Placebo | Placebo/CBTsh | Sibutramine/CBTsh | Total
Number analyzed (Participants) | 26 | 27 | 25 | 26 | 104
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.2 (10.3) | 43.2 (12.4) | 45.7 (12.4) | 45.6 (9.4) | 44.2 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 18 | 20 | 16 | 73
  Male | 7 | 9 | 5 | 10 | 31
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 13 | 12 | 12 | 10 | 47
  African-American | 8 | 12 | 6 | 10 | 36
  Hispanic-American | 4 | 2 | 4 | 4 | 14
  Other | 1 | 1 | 3 | 2 | 7
Age at onset of Binge Eating Disorder (BED) [Mean (Standard Deviation); unit: years] | 25.7 (11.2) | 25.5 (11.1) | 25.7 (15.1) | 29.1 (13.1) | 26.2 (12.5)

OUTCOME MEASURES:

1. Primary Outcome: Binge Eating (Remission)
Description: Remission from binge eating (zero binge episodes during previous 28 days)
Time Frame: 4 months treatment; 6 and 12 month follow up post treatment
Measure: Number; unit: participants
Arm/Group | Sibutramine | Placebo | Placebo/CBTsh | Sibutramine/CBTsh
Number analyzed (Participants) | 26 | 27 | 25 | 26
participants
  Remission at Post-treatment | 10 (11.4) | 8 (9.9) | 6 (7.6) | 6 (8.0)
  Remission at 6 month follow up | 5 | 11 | 10 | 13
  Remission at 12 month follow up | 5 | 10 | 10 | 11
Statistical Analysis 1: Comparison: Sibutramine vs Placebo vs Placebo/CBTsh vs Sibutramine/CBTsh; Post-treatment; Test type: Superiority or Other; p = 0.60, Chi-squared; df=3
Statistical Analysis 2: Comparison: Sibutramine vs Placebo vs Placebo/CBTsh vs Sibutramine/CBTsh; 6 month follow up; Test type: Superiority or Other; p = 0.13, Chi-squared; df=3
Statistical Analysis 3: Comparison: Sibutramine vs Placebo vs Placebo/CBTsh vs Sibutramine/CBTsh; 12 month follow up; Test type: Superiority or Other; p = 0.29, Chi-squared; df=3

2. Primary Outcome: BMI
Description: BMI (kg/m^2) was measured 4 months after treatment.
Time Frame: 4 months
Population: Participants with complete data reported here (i.e., no imputation)
Measure: Mean (Standard Deviation); unit: BMI (kg/m^2)
Arm/Group | Sibutramine | Placebo | Placebo/CBTsh | Sibutramine/CBTsh
Number analyzed (Participants) | 21 | 19 | 22 | 22
BMI (kg/m^2) | 38.4 (7.2) | 39.6 (5.7) | 35.9 (5.6) | 35.6 (4.6)

ADVERSE EVENTS:
Arm/Group | Sibutramine | Placebo | Placebo/CBTsh | Sibutramine/CBTsh
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/27 | 0/25 | 0/26
Other Adverse Events (participants affected / at risk) | 1/26 | 2/27 | 0/25 | 1/26
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sibutramine (N=26) | Placebo (N=27) | Placebo/CBTsh (N=25) | Sibutramine/CBTsh (N=26)
Elevated blood pressure (Vascular disorders) | 1 | 2 | 0 | 1 — Patients medically withdrawn due to elevation in blood pressure during treatment (i.e., in excess of 145/90 BP, 100 pulse)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes